CLINICAL TRIAL: NCT06936930
Title: A Study on Reproductive and Psychological Health in Aplastic Anemia Patients
Brief Title: Reproductive and Mental Health of Patients With Aplastic Anemia
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: QTJC2025034
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-04

CONDITIONS: Aplastic Anemia; Reproductive Health
Keywords: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Female group: To evaluate the reproductive health and psychological status of reproductive-age patients with aplastic anemia and to monitor long-term changes in sex hormone levels under different treatment regimens.
  Interventions: Other: Sex hormone monitoring
- Male group: To evaluate the reproductive health and psychological status of reproductive-age patients with aplastic anemia and to monitor long-term changes in sex hormone levels under different treatment regimens.
  Interventions: Other: Sex hormone monitoring

INTERVENTIONS:
Other: Sex hormone monitoring — Sex hormone monitoring includes the concentrations of follicle-stimulating hormone (FSH), luteinizing hormone (LH), estradiol (E2), progesterone (P), prolactin (PRL), and testosterone (T).

SUMMARY:
Aplastic anemia (AA) is a hematological disease characterized by bone marrow failure, leading to varying degrees of anemia, leukopenia, and thrombocytopenia. With the advancement of immunosuppressive therapy and hematopoietic stem cell transplantation, the survival of AA patients has significantly improved. However, these treatment approaches may result in reproductive system impairment.

Reproductive health has been a major concern among reproductive-age AA patients. In female patients, it often manifests as irregular menstruation, amenorrhea, and infertility; while in male patients, it may present as reduced sperm count and low sperm motility. The reproductive impairment observed in AA patients may be attributed to various factors, including the disease's underlying pathophysiology, side effects of used medications such as androgens and the toxicity conditioning agents during transplantation.

Notably, immunosuppressive agents (such as cyclosporine and antithymocyte globulin) and chemotherapeutic drugs (such as cyclophosphamide) can suppress hematopoiesis and directly damage the gonads, thereby impairing reproductive function. Furthermore, long-term use of these medications may disrupt the endocrine system, affecting the secretion of sex hormones and overall reproductive capacity. Additionally, chronic anemia in AA patients can lead to compensatory physiological changes in other body systems, which may also indirectly affect reproductive health.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AA
* Male or female, aged 18-40 years
* ECOG performance status ≤2
* Willing and able to comply with the requirements for this study and written informed consent

Exclusion Criteria:

* Diagnosis of inherited bone marrow failure syndromes
* Combined with other hematological diseases
* Chemotherapy-induced bone marrow failure
* Pregnant or breastfeeding women
* Subjects with a history of mental illness or severe psychological disorders
* Subjects with a history of reproductive system cancer (eg, penile cancer, testicular cancer, prostate cancer, ovarian cancer, cervical cancer, vaginal cancer, etc.)
* Subjects that the investigator believes have other reasons that make them unsuitable for inclusion in this study

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: 300 Reproductive-age males and 300 females diagnosed with acquired aplastic anemia.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with abnormal sex hormone levels | Baseline, 6 months post-treatment, 12 months post-treatment
  The concentrations of FSH, LH, E2, P, PRL and T.

SECONDARY OUTCOMES:
Stress levels | Baseline
  Perceived Stress Scale (PSS-10) can range from 0 to 40 with higher scores indicating higher perceived stress.
Depression symptoms | Baseline
  Patient Health Questionnaire (PHQ-9) can range from 0 to 27 with higher scores indicating greater severity of depression.
Social support | Baseline
  Medical outcomes study social support survey (MOS-SSS) can range from 0 to 100 with higher scores indicate greater perceived social support.

CONTACTS AND LOCATIONS:
Locations (1):
- Regenerative Medicine Center, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No